CLINICAL TRIAL: NCT00444093
Title: Prospective Randomized Open Label Study of the Treatment of Therapy-associated Diarrhea During Percutaneous Radiation Therapy of the Small Pelvis. - Comparison of Loperamide and Tincture of Opium
Brief Title: Prospective Randomized Open Label Study of the Treatment of Therapy-associated Diarrhea During Percutaneous Radiation Therapy of the Small Pelvis. - Comparison of Loperamide and Tincture of Opium -
Acronym: Loop
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: bad recruitment
Sponsor: Philipps University Marburg (Other)
Collaborators: Maros Arznei GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-002948-28; KKS-73-05
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2018-04

CONDITIONS: Diarrhea; Enteritis; Cancer
Keywords: radiation therapy; diarrhea; enteritis; supportive therapy; therapy associated diarrhea; therapy associated enteritis; radiation therapy of the small pelvis
MeSH Terms: conditions — Diarrhea; Enteritis; Neoplasms

STUDY DESIGN:
Intervention Model Description: Comparision between treatment with Tinctura Opii normata and Loperamid in patients with therapy-associated diarrhea during radiaton therapy of small pelvis
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Opii normata treatment (Experimental): Treamtment with opii normata in case of diarrhea
  Interventions: Drug: Opii normata treatment
- Loperamid Treatment (Experimental): Treatment with Loperamid in case of diarrhea
  Interventions: Drug: Loperamid Treatment

INTERVENTIONS:
Drug: Opii normata treatment — After beginning of diarrhea grade 1:
  5 drops tincture of opium three times a day
  After beginning of diarrhea grade 2:
  Intensive therapy with 15 drops tincture of opium three times a day.
  Arms: Opii normata treatment
Drug: Loperamid Treatment — All patients who receive as a result of randomisation loperamide
  After beginning of diarrhea grade 1:
  Initial 4mg and 2mg after any unformed stool. The maximum dose amounts to16mg per day.
  After beginning of diarrhea grade 2:
  Intensive therapy with 2mg loperamide every 2 h. The maximum dose amounts to 16mg per day.
  Arms: Loperamid Treatment

SUMMARY:
Therapy-associated diarrhea during radiation therapy of small pelvis (including enteritis as a result of radiation therapy and enteritis as a result of radiation- and chemotherapy) is a common problem in multimodal cancer therapy. We investigate the therapeutic effect of either loperamide or tinctura opii in therapy- associated diarrhea in patients who receive radiation therapy of the small pelvis with or without chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who will undergo a percutaneous radiation therapy in the area of the small pelvis. This includes patients with following malignancies: rectal carcinoma, prostate carcinoma, endometrial carcinoma, cervix carcinoma.
* Diarrhea grade 1 and grade 2 (Classification NCI-CTCAE Version 3.0)
* ECOG-Grade 0-2
* Enlightenment and written declaration of consent to the participation.

Exclusion Criteria:

* Pregnant patients or patients in lactation period.
* Severe dysfunction of liver or kidneys
* Injury or illness of brain e.g. increased intracranial pressure, cerebral arteriosclerosis
* Epilepsy
* Hypersensitivity to components of loperamide or tincture of opium
* Ileus
* Toxic megacolon
* Pseudomembranous colitis/ antibiotic-associated colitis
* Diarrhea associated with fever and bloody stools
* Acute increase of colitis ulcerous or bacterial colitis caused by invasive pathogenes
* Severe respiratory dysfunction or severely limited lung function e.g. bronchial asthma, bronchitis
* Dysfunctional draining of biliary area, biliary colics.
* Concomitant or earlier addiction of alcohol or opiates
* Severe heart disease
* Pheochromocytoma
* Acute hepatic porphyria
* Cor pulmonale
* Morbus Addison
* Severe hypothyroidism
* Organisational problems or circumstances which prevent a complete collection of required data
* Artificial anus
* Participation in a clinical trial within the last 30 days before involvement
* Participation in an other clinical trial at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-03-05 (Actual); Primary Completion 2008-02-29 (Actual); Study Completion 2008-02-29 (Actual)

PRIMARY OUTCOMES:
Treatment Efficacy | 90 days
  In this study efficacy of loperamide and tincture of opium is linked to the respective proportions of patients where diarrhoea of grade > 2 is successfully averted during (cancer) therapy.

SECONDARY OUTCOMES:
Quality of life EORTC-QLQ C30 | 90 days
  Quality of life will be assessed with the EORTC-QLQ C30 questionnaire
Diarrhea Assessment | 90 days
  The quality and quantity of diarrhea will be assessed with a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bieker, MD, Principal Investigator — center of radiology, departement of radiation therapy, clinical center Giessen and Marburg